CLINICAL TRIAL: NCT03384407
Title: Measurement of the Recovery and Lifespan of Red Blood Cells From Pathogen-Reduced, Stored Blood Units Using Cellular Biotinylation
Brief Title: Recovery and Lifespan of Red Blood Cells From Pathogen-reduced, Stored Blood Units
Acronym: BIO-CR-RBC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cincinnati (Other)
Collaborators: Cerus Corporation (Industry); Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jose Cancelas, Professor, Research Division Director, Hoxworth Blood Center, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2018-01
Record Dates: First submitted 2017-12-19; First posted 2017-12-27 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Red Cell Survival in Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Open label (Experimental): Red cell recovery/survival analysis of untreated and INTERCEPT treated RBC concomitantly
  Interventions: Device: Red cell survival in INTERCEPT treated red cells

INTERVENTIONS:
Device: Red cell survival in INTERCEPT treated red cells — Red cell recovery/survival analysis of untreated and INTERCEPT treated RBC concomitantly

SUMMARY:
The pilot study has two objectives: 1) to assess the post-infusion viability of INTERCEPT RBC by measuring the 24 hour post-infusion recovery ("PTR24") and lifespan of autologous RBCs prepared with the INTERCEPT System for RBC after storage for 35 days under standard blood banking conditions using two different RBC labels; 51-chromium and biotin. The control will be conventional untreated RBCs stored for 35 days; and 2) comparison and contrast of PTR24 and lifespan results of the 51-chromium and biotin labeling methods of RBC stored for 35 days under standard blood banking conditions. The purpose of gathering these data is to obtain more meaningful survival data for stored conventional and INTERCEPT RBCs over the entire 120 d RBC lifespan (51-Cr labeled RBC permits a maximum 28 d assessment as a result of 51-Cr's variable, progressive elution from RBC and radioactive half-life).

DETAILED DESCRIPTION:
Each subject will receive one infusion of autologous, radiolabeled and BioRBC labeled INTERCEPT RBCs (Test RBCs) and one infusion of autologous BioRBC labeled untreated RBCs (Control RBCs) concomitantly. Each infusion will be approximately 20 mL, i.e., 10 mL of 51-chromium labeled RBC, and 10 mL of either BioRBC-6 or BioRBC-18 which will be stratified as indicated above based on the Test or Control designation.

Treatment Compliance Healthy subjects who understand the study commitments and sign the informed consent will be enrolled in the study. Treatment compliance and follow-up testing will be tracked by the Investigator, recorded on the case report form (CRF), and monitored by the Sponsor.

ASSESSMENT OF EFFICACY

Efficacy Parameters

Efficacy endpoints include the following:

Primary Efficacy Endpoint(24)

- 24 hour post-infusion recovery of autologous RBC stored in AS-5 for 35 days and then labeled with either 51Cr or biotin.

Secondary Efficacy Endpoints(25)

* Mean lifespan of autologous RBC stored for 35 days and then labeled with either 51Cr or biotin
* Median lifespan (T50) of autologous RBC stored for 35 days and then labeled with either 51Cr or biotin
* Area under the curve (AUC) determined using data points collected forRBC lifespan of autologous, radiolabeled or BioRBCs

  e) Dose determination and duration

Methods and Timing of Efficacy Parameters This study consists of a single treatment period where Control biotinylated (using a RBC surface density of 6 or 18 mcg of sulfo-NHS-biotin per mL RBC) are administered, i.e., co-infused at a single point in time with Test INTERCEPT-treated biotinylated RBC (using a concentration of 18 or 6 mcg of sulfo-NHS-biotin per mL RBC) and INTERCEPT-treated, radiolabeled (51Cr) RBC. All 6 subjects will receive both control and S-303-treated (test) RBCs concomitantly and the only difference between the two sets of 3 subjects will be the level of biotinylation of the control or test RBC.

The study is stratified and control or test RBC will be labeled alternatively with either 6 or 18 mcg of sulfo-NHS-biotin per mL RBC. RBC from three individuals (subjects 1, 3 and 5) will be labeled with 6 and 18 mcg of sulfo-NHS-biotin per mL RBC for control and test RBC, respectively. Other three individuals (subjects 2, 4 and 6) will be labeled with 6 and 18 mcg of sulfo-NHS-biotin per mL RBC for Control and Test RBC, respectively. The objective of this stratification is to ensure that no bias is introduced by the biotin label density into one of the arms of the study.

f) Description of observations and measurements

On Day 0 of each treatment period the subject will donate two units of packed RBC (double RBC automatized donation, Trima - Terumo BCT apheresis system); the units will be leukocyte reduced by in-line filtration and the RBC concentrates will be prepared in additive solution (AS-5).

One of the two units will be stored immediately at 1-6ºC for 35 days (Control unit). This conventional RBC component represents the Control RBCs in this study.

The Test RBC unit will be prepared by processing using the INTERCEPT Blood System for Red Blood Cells. In vitro biochemical and morphological parameters of the study RBC components (Table 1) will be measured on Day 0 after preparation of RBC concentrates in AS-5 (prior to study treatment), post processing and prior to storage (Test only), and again on Day 35 (prior to infusion back in to study subjects) to evaluate the RBC quality of the processed/stored RBC units. The data collected for the in vitro characteristics will be summarized using descriptive statistics.

Table 1. Biochemical parameters analyzed on day 0 and day 35 of storage of control- and treated RBC units.

Parameter Hb content/unit Hemolysis pH pO2 pCO2 Glucose (extracellular) Lactate (extracellular) Bicarbonate (extracellular) Sodium (extracellular) Potassium (extracellular)

On Day 35 of RBC storage each treatment period, an aliquot of Control RBCs will be biotinylated (6 or 18 mcg/mL). From the Test unit, two aliquots will be drawn; the first aliquot will be radiolabeled with 51Cr and the second aliquot will be biotinylated at 6 or 18 mcg/mL. Re-infusion of the two biotinylated autologous RBC (Control and Test) specimens along with the 51Cr labeled autologous RBC (Test) will measure recovery and survival (approximately total: 20 mcCi). Also on Day 35, a 20 mL sample of fresh blood will be drawn from the subject and the RBCs labeled with 99mTc and Bio-54. Re-infusion of the fresh 99mTc RBC and fresh Bio-54 will allow determination of subject blood volume or number of circulating RBC.

Five types of RBC will be mixed and infused: a) fresh RBC labeled with 99mTc and BioRBC-54; b) fresh Bio-54 labeled RBC; c) Stored, Control or Test RBC biotinylated at density 6 mcg/mL; d) Stored, Test or Control RBC biotinylated at density 18 mcg/mL; and, e) Stored, Test, RBC labeled with 51Cr. All aliquots will be labeled separately and mixed for a volume of ~50 mL. The 50 mL of autologous RBCs will be infused through a peripheral vein using an 18-19 gauge butterfly needle (at an approximate rate of 5 mL/min).

Blood samples, from the subject's contralateral arm, will be collected immediately pre-infusion and at 5, 7.5, 10, 12.5, 15, 20, 30 minutes and 24 hours after completion of the infusion to permit extrapolation to T=0 for 51Cr determination of blood volume as previously published by our group (16, 17, 26-30).

Additional blood samples will be collected at 48 and 72 hours and 7 days post-infusion, and then weekly through 28 days (days 37, 38, 42, 49, 56 and 63 post-infusion) and bi-weekly from then on (days 77, 91, 105, 119, 133, 147). After collection of the final blood sample in Treatment Period 2, subjects will be discharged from the study.

Upon completion of the study, each of the 6 subjects will have provided 2 units of whole blood and receive 1 infusion of autologous radiolabeled Test or Control RBCs and 1 infusion of autologous radiolabeled Control or Test RBCs.

The study assessments used to evaluate both efficacy and safety are presented below (Section 1).

g) Clinical procedures, laboratory tests, monitoring drug effects and minimizing risks

Section 1: Study Assessments and data collection Screening: Day -28 to 0

* Explain study to subject
* Obtain signed Informed Consent
* Medical history
* Blood donor physical exam
* Vital signs
* Concomitant medications, i.e., other than those excluded
* Samples for laboratory tests: Hematology, serum Chemistry, and Blood Donor testing (microbiological, ABO/Rh) screening panel (following FDA/AABB requirements).
* Direct and Indirect Antiglobulin Test (DAT/IAT)
* ABO and Rh type (part of the donor panel)
* Serum or plasma sample to test for antibody specific to INTERCEPT RBC and antibody specific to biotinylated RBC
* Stratify subjects to receive BioRBC-6 or BioRBC-18 for INTERCEPT treated RBCs
* Serum or plasma sample for iron status testing: ferritin (being acceptable, ferritin > 26 ng/mL) Prior to Blood Collection, Day 0
* Intercurrent illness
* Vital signs
* Concomitant medications
* Hemoglobin/hematocrit

Double RBC Collection, Day 0 Trima Collection Procedure Parameters and Schedule (AC Ratio, etc.)

1. Anticoagulant (AC) ratio The AC ratio is a parameter that is configurable on the Trima System. The red cells units will be collected at a whole blood to anticoagulant ratio of 11.
2. Run time The run time will be limited to a maximum of 120 minutes. Double RBC products will be collected when using the Trima RBC, Plasma sets and are expected to take approximately 30 minutes total.

   RBC Component - Prior to Study Treatment Day 0

   - Collect sample from the study Control and Test RBC units for in vitro lab assessments

   RBC Component - Study Treatment, Day 0-1
   * Process and/or perform INTERCEPT Process for RBCs in one of the two donated blood units.
   * Collect a sample from the Test RBC component (in vitro assessments)
   * Place Control and Test RBC components in traditional blood bank storage (1-6ºC).

   Post Blood Collection, Day 1 (24±6 hours post donation)
   * Concomitant medications
   * Intercurrent illness
   * Collect AEs and SAEs (Note: These data may be collected by phone)

   RADIOLABELING, BIOTINYLATION AND RE-INFUSION OF AUTOLOGOUS RBC ALIQUOTS Prior to Re-Infusion of autologous labeled, Day 35 (within 6 hours prior to infusion)
   * Collect a fresh 20 mL sample of subject's blood for 99mTc and BioRBC-54 labeling
   * ABO type
   * Confirm the identity of the RBC study component by clerical analysis of chain-of-custody documentation and blood bag labels following industry standards and AABB/FDA regulations
   * Samples for laboratory tests: Hematology and serum chemistry
   * Pregnancy test (if female subject)
   * Serum or plasma samples for INTERCEPT antibodies RBC and anti-BioRBC antibodies
   * Samples for RBC recovery, mass, lifespan
   * Intercurrent illness
   * Vital signs
   * Height and weight
   * Concomitant medications
   * Collect AEs and SAEs since donation.

   RBC Component:

   Prior to Infusion, Day 35

   - Label 10 mL aliquot of 35 day-old study RBC with 51Cr
   * Label fresh 10 mL aliquot of subject's RBC with 99mTc and BioRBC-54
   * Collect a sample of study RBC component (for in vitro assessments)

   Infusion of Autologous Study RBCs, Day 35

   - Infusion of a mixture of five ~10 mL (total ~50 mL) aliquots of autologous blood (all mixed together and infused at rate of 5-7 mL/min) including: a) fresh RBC labeled with 99mTc and BioRBC-54; b) fresh Bio-54 labeled RBC; c) Stored, Control or Test RBC biotinylated at density 6 mcg/mL; d) Stored, Test or Control RBC biotinylated at density 18 mcg/mL; and, e) Stored, Test, RBC labeled with 51Cr. All aliquots will be labeled separately and mixed for a volume of ~50 mL. The 50 mL of autologous RBCs will be infused through a peripheral vein using an 18-19 gauge butterfly needle (at an approximate rate of 5 mL/min). (Note: The remainder of the two 35 day-old INTERCEPT treated and non-treated Control RBC units are discarded.)
   * Concomitant medications
   * Collect AEs and SAEs

     * Hematology tests: CBC including hemoglobin, hematocrit, platelets, MCV, MCH, MCHC, RDW ** Serum chemistry tests: calcium, bicarbonate, chloride, inorganic phosphate, potassium, sodium, cholesterol, glucose, total protein, triglycerides, LDH, ALT, AST, total bilirubin, BUN, & creatinine.

       * Includes: serum or plasma ferritin, iron, iron binding capacity, transferrin saturation † Vital signs: heart rate, respiratory rate, blood pressure and temperature. If fever within 24 hours of infusion (temperature>39°C or >38˚C with shaking chills) culture the subject and the RBC bag.

   The assessments and data collection beginning the day following the RBC infusion until Study Day 147 (day 112 post-infusion) are shown in the Table 1.

   ASSESSMENT OF SAFETY The timing of study safety assessments is presented in the Table.

   Safety Parameters

   Safety endpoints include the following:

   Primary Safety Endpoint
   * Incidence of antibody specific to INTERCEPT treated RBCs
   * Incidence of antibody specific to biotinylated RBCs Secondary Safety Endpoint
   * Incidence of adverse and severe adverse events as described below in the section titled, "Recording and Reporting Adverse Events." The INTERCEPT Treatment System medical device will be monitored for device deficiencies, including malfunctions and adverse device effects.

   Methods and Timing of Safety Parameters In this study, the Sponsor/Investigator, J.A. Cancelas, will collect and record adverse events (AEs) for 24 hours following collection of each whole blood unit and for 24 hours following each infusion of study RBCs. Serious adverse events (SAE) will be collected and recorded from the time the first unit of whole blood is collected until the completion of the study (Table).

   Subjects will be actively monitored for AEs during blood collection and during the study RBC infusions, and until they are discharged. After discharge, all AEs reported to the qualified study staff will be recorded. AE and SAE data may be collected by phone or in person by study staff. Vital signs are collected prior to and following each study infusion. In the event that a subject develops within 24 hours after a study RBC transfusion post-infusion fever, defined as a temperature >39°C or a temperature >38°C with shaking chills (rigors) or signs and symptoms consistent with bacterial sepsis, the subject's blood will be cultured and the Blood Center will be notified to culture the RBCs remaining in a segment or the residual Test or Control RBC components.

   Our group will test subject serum or plasma for antibody specific to INTERCEPT RBCs and BioRBC; these samples will be obtained from each subject pre-infusion, 14 days after infusion, and 28 days after infusion and monthly thereafter to study day 147 (see Table). If an antibody specific to INTERCEPT treated RBCs is identified, samples will be sent to an independent laboratory for confirmation (the UCLA/American Red Cross, Pomona). Blood samples for hematology and chemistry panels will be obtained from each subject Study Days: pre-infusion (day 35), 24 hours after the infusion (day 36), 56 days after infusion (day 91) and 112 days after infusion (day 147, at the end of the study). Clinically significant laboratory findings will be recorded as adverse events. The laboratory assessments are identified in the Table 1.

   Transfusion Reactions Although transfusion reactions are unlikely due to the small infusion volume, clinically significant transfusion reactions will be recorded as adverse events.

   Suspected Transfusion Related Sepsis Subjects will be monitored for infusion-related adverse events including infusion-related sepsis following the study infusion. To provide an unaltered sample of the blood infusate aliquot transfused into a subject, the remainder of this aliquot will be sent for bacterial culture.

   In the event that a subject develops post-infusion fever, defined as a temperature >39°C or a temperature >38°C with shaking chills (rigors) or signs and symptoms consistent with bacterial sepsis within 24 hours after a study RBC infusion, the subject's blood will be cultured and the remaining stored component will be cultured.

   Cultures will be performed by investigators at the Hoxworth Blood Center according to standard operating procedures at the Hoxworth Blood Center. If bacteria are recovered from both the patient's blood and the RBC component, samples of the isolates will be sent to the University of Cincinnati Hospital laboratory to determine if the recovered organisms are identical. Infusion-induced sepsis will not be established unless the same organism(s) is recovered from both the RBC component and from the study subject.

   Detection and Confirmation of Antibody Specific to INTERCEPT RBCs Although not anticipated to occur in this study due to the limited exposure to Test RBC, all subjects will be tested for the presence of antibody specific to INTERCEPT treated RBC at study entry (naturally occurring antibody) and at specified times during the study (Table 1).

   The presence of antibody will be evaluated using a formally validated gel card IAT that is routinely used in many blood centers for transfusion compatibility testing in conjunction with a panel of frozen reagent INTERCEPT RBCs. The frozen RBC screening panel is composed of reagent RBCs from 3 specifically phenotyped blood group O donors, and is analogous to routine antibody screening panels used in regular blood banking practice. Each cell in the panel of 3 consists of untreated RBCs, cells carrying a "high" level of acridine adducts and cells carrying a "low" level of acridine adducts. The screening panel was designed as a sensitive screening test for the presence of INTERCEPT RBC antibodies in the presence of most common alloantibodies. Gel card agglutination will be scored 1+ to 4+ based on manufacturer's recommendation.

   For result interpretation, if the RBC screening panel score is positive with 3/3 of the INTERCEPT RBCs carrying either 'high" and/or "low" levels of acridine adducts AND with 0/3 with the corresponding Control untreated RBCs the sample is classified as "reactive for INTERCEPT RBC antibodies.

   Antibody confirmation and characterization will be performed at the ARC Immunohematology Reference Laboratory, Pomona and will include acridine specificity by agglutination inhibition (neutralization) using a soluble acridine analog of amustaline, antibody titer, antibody isotype and thermal amplitude.

   If the presence of antibody specific to INTERCEPT RBC is established, this does not determine whether that antibody is physiologically active or clinically significant, this can only be determined by any one of the following criteria indicative of accelerated RBC clearance in the absence of active bleeding, organ-mediated RBC sequestration, severe erythroid hypoplasia or other concurrent medical cause for acute anemia not associated with transfusion.

   Detection and Confirmation of Antibody Specific to BioRBC As with INTERCEPT RBCs, subjects will be screened prior to transfusion for the presence of naturally occurring or pre-existing antibody to BioRBC (18). This will be done using the same gel card agglutination as for the INTERCEPT RBCs but using BioRBCs incubated with subject serum or plasma. Briefly, 50 µL of 0.8% hematocrit target BioRBC-N or unlabeled RBC will be prepared from a blood GpO donor and added to the gel column. Subject plasma (25 µL) is added to the target RBCs and incubated at 37˚C for 30 min. Gel cards are subsequently centrifuged for 10 min. The presence of BioRBC agglutination is quantified using the manufacturer's gradation-specific definitions of reactivity. Reactivity scores will be based on manufacturers recommendation 0-4+ but, in addition, a score of 1+ (i.e., agglutination in lower half of matrix) will be further sub-classified into three increasingly reactive 1+ designations: 1) ± indicates a slanted pellet with a few agglutinated RBC; 2) 1w indicates a slanted pellet with more agglutinated RBC; and 3) 1+ indicates a disrupted RBC pellet with more agglutinated cells. As with the detection of INTERCEPT-specific antibodies, the detection of specific antibodies to BioRBC does not determine whether that these antibodies are physiologically active or clinically significant.

   Confirmatory testing of the induction of BioRBC-induced antibodies will be performed by agglutination inhibition (neutralization) with biotin compounds, e.g., biocytin, biotinylated gelatin or biotinylated albumin is able, are able to neutralize anti-BioRBC antibodies. So far, all identified preexisting, naturally occurring anti-BioRBC antibodies are neutralized by biotin compounds, while the induced anti-BioRBC antibodies are expected to be inhibited by BioRBC and not by free biotin as previously published by our group (5).

   Recording and Reporting Adverse Events Adverse Event Definition An AE is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the medicinal product (in this study BioRBC and INTERCEPT RBC) whether or not related to the medicinal product (International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH-E2A, section 2.1)

   Serious Adverse Event Definition

   Some AEs are considered "serious" when the outcome of the event poses a threat to a patient's life or functional status. A serious adverse event (SAE) is an AE that results in the following outcomes:
   * Results in death
   * Life-threatening
   * Requires inpatient hospitalization or prolongation of existing hospitalization
   * Results in persistent or significant disability/incapacity
   * Is a congenital anomaly/birth defect
   * Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the subject and/or may require intervention to prevent one of the outcomes listed in this definition (ICH E2A section II/B).

   Adverse Device Effect Definition An Adverse Device Effect (ADE) is defined as an adverse event related to the use of an investigation medical device.

   Unanticipated Adverse Effect Definition An unanticipated adverse effect (UAE) is defined as any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, the process, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan or application (including a supplementary plan or application), or any other unanticipated serious problem associated with a device that relates to the rights, safety, or welfare of subjects (21 CFR 812.3).

   Reporting Adverse Events AEs will be documented on the appropriate case report form (CRF), regardless of whether or not they are classified as associated with the study product.

   If an AE meets the criteria of a serious adverse event (SAE) or unanticipated adverse device effect (UAE) as described above, the Sponsor/PI will halt the study and notify the FDA within 7 days.

   The Investigators will comply with the applicable regulatory requirement(s) related to the reporting of serious adverse events to the IRB. An Investigator shall submit to the Sponsor and to the reviewing IRB a report of any unanticipated adverse device effect occurring during an investigation as soon as possible, but in no event later than 10 working days after the Investigator first learns of the effect.

   The Sponsor will report suspected unexpected serious adverse reactions and/or unanticipated adverse device effects to comply with the applicable regulatory requirement(s).

   Assessing Seriousness and Severity of an Adverse Event The Investigator is required to assess if the adverse event is non-serious or serious, the latter is defined as an event that resulted in any of the following outcomes: death, a life-threatening event (results in an immediate risk of death from the reaction as it occurred), inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant disability/incapacity, a congenital anomaly/birth defect, or another important medical event.

   The term "severe" is used to describe the intensity (severity) of a specific event (as in mild, moderate, or severe); the event itself, however, may be of relatively minor medical significance (such as severe headache). Severity is not the same as "serious", which is based on patient/event outcome or treatment criteria associated with events that pose a threat to a patient's life or functional status.

   Seriousness (not severity) serves as a guide for defining regulatory reporting obligations. The National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE, version 4.03) is used to assess and classify the intensity/severity of an event.

   Assessing Causal Relationship of an Adverse Events The Investigator will assess whether there is a reasonable possibility that the study blood collection or RBC infusion caused or contributed to an adverse event.

   Determination of whether there is a reasonable possibility that the study RBC component caused or contributed to an adverse event includes assessing temporal relationships, biologic plausibility, dechallenge/rechallenge information (if available), association (or lack of association) with underlying disease, and presence (or absence) of a more likely cause.

   The scale for assessing the causal relationship of an adverse event to the study RBC component (imputability levels) follows:

   Causality Assessment Scale Imputability Level Explanation Excluded When there is conclusive evidence beyond reasonable doubt for attributing the adverse event to alternative causes. Unlikely When the evidence is clearly in favor of attributing the adverse event to causes other than the study RBC component.
   1. Possible: When the evidence is indeterminate for attributing adverse event either to the RBC component or to alternative causes.
   2. Likely: Probable When the evidence is clearly in favor of attributing the adverse event to the RBC component.
   3. Certain: When there is conclusive evidence beyond reasonable doubt for attributing the adverse event to the RBC component.

   Assessing Intensity of an Adverse Events The Investigator is required to assess the intensity (severity) of each adverse event using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE)

   Adverse Event Follow up All SAEs will be followed until resolution, or the Investigator judges the event to be chronic or stable.

   Stopping Rules

   The following SR will be applied to all study subjects throughout the trial whenever this study's sponsor/PI (José Cancelas, M.D., Ph.D.,) and/or Clinical Monitor (Patricia Carey MD, Professor of Pathology, Medical Director, Hoxworth Blood Center)) agree that any of the following have occurred:
   1. An SAE that is determined to be possibly, probably, or definitely related to the infusion of autologous BioRBC;
   2. An AE related to the infusion of autologous BioRBC jeopardizes the subject's health or safety;
   3. An AE requiring medical or surgical intervention related to the infusion of autologous BioRBC is required to prevent occurrence of an SAE;
   4. A post-infusion of hemolysis event as assessed by anti-BioRBC antibody detection using the IgG gel card assay developed by our group.

   If any of the above conditions occur, the study will be paused and reported to FDA and IRB as required by current regulations to assess continuation of the study. Infused subjects will remain being followed as long as needed to identify the consequences of the AEs identified. Since there are no additional experimental BioRBC transfusions administered as part of this study, "continuation of the study" is understood to mean a continuation of the monitoring of biologic samples as already outlined in this study, but possibly including other testing as deemed appropriate by the study's sponsor/PI, Clinical Monitor, FDA and/or IRB.

ELIGIBILITY:
Subject Inclusion Criteria

* Up to 12 subjects will be enrolled for a maximum of 6 eligible subjects in the pilot study to provide preliminary RBC survival data to support a subsequent adequately powered study capable of addressing the two objectives as stated above.
* Age ≥18 years, of either gender
* Normal health status (as determined by the Investigator review of medical history and blood donor physical exam)
* Weight over 140 lbs.
* Complete blood count (CBC; including RBC indices MCV, MCH, MCHC, and RDW) and serum chemistry values within normal limits (including calcium, bicarbonate, chloride, inorganic phosphate, potassium, sodium, cholesterol, glucose, total protein, triglycerides, LDH, ALT, AST,total bilirubin, BUN, creatinine). Values outside of normal reference range if considered not to be clinically significant may be allowed with a protocol exception.
* Minimum hemoglobin levels of 13 g/dL for female and 14 g/dL for male subjects
* Negative blood donor screening test panel for HIV, HBV, HCV, HTLV, Syphilis, WNV and Zika virus
* Female subjects of childbearing potential and male subjects must agree to use a medically acceptable method of contraception throughout the study periods. A barrier method of contraception must be included, regardless of other methods.
* Meet or exceed AABB guidelines for blood donation (with the exception of travel deferrals).
* Signed and dated informed consent form

Subject Exclusion Criteria

* Clinically significant acute or chronic disease (as determined by the Investigator)
* History of RBC autoantibodies/autoimmune hemolytic anemia, RBC alloantibodies or autoimmune disease
* History of congenital red cell disorders including glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Positive Direct (DAT) and Indirect antiglobulin test (IAT)at study entry
* Immunosuppressive therapy (e.g., oral or IV prednisone) within the past 28 days
* Treatment with any medication known to affect RBC viability
* Pregnant or nursing female
* Male subjects or female subjects of childbearing potential not using effective contraception
* Participation in another clinical study currently or within the past 28 days
* Prior exposure to INTERCEPT treated or BioRBCs
* Pre-existing antibody specific to INTERCEPT RBCs or BioRBC
* Subjects are excluded if receiving immunosuppressive therapies (e.g., oral or intravenous corticosteroids) due to their potential to obscure immunogenicity or immunoreactivity to Test RBCs.
* Subjects donating blood for any other purpose
* Subjects who have received blood transfusion within the previous year
* Subjects who are enrolled in another study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
24 hour post-infusion recovery of autologous RBC stored in AS-5 for 35 days and then labeled with either 51Cr or biotin. | 24 hours

SECONDARY OUTCOMES:
Mean lifespan of autologous RBC stored for 35 days and then labeled with either 51Cr or biotin | days 37, 38, 42, 49, 56, 63, 77, 91, 105, 119, 133 and 147
Median lifespan (T50) of autologous RBC stored for 35 days and then labeled with either 51Cr or biotin | days 37, 38, 42, 49, 56, 63, 77, 91, 105, 119, 133 and 147
Area under the curve (AUC) determined using data points collected for RBC lifespan of autologous, radiolabeled or BioRBCs | days 37, 38, 42, 49, 56, 63, 77, 91, 105, 119, 133 and 147

CONTACTS AND LOCATIONS:
Locations (1):
- Hoxworth Blood Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided